CLINICAL TRIAL: NCT05365334
Title: Skeletal Muscle and Adipose Tissue Responses After Acute Exercise: Comparing Effects of Three Different Intensities
Acronym: 3X
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Professor of Movement Science and Director of the Substrate Metabolism Laboratory (SML) at the University of Michigan School of Kinesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00204857
Record Dates: First submitted 2022-04-08; First posted 2022-05-09 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Cellular Responses Within Skeletal Muscle in Response to Exercise of Different Intensities; Relationship Between the Cellular Responses in Skeletal Muscle and the Changes in the Metabolomic Profile; Changes Within Adipose Tissue in Response to Exercise at the Three Different Intensities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low-intensity continuous exercise (Experimental): subjects will exercise at 30% maximal oxygen consumption (VO2max) for 45-60 minutes
  Interventions: Behavioral: Low intensity exercise session
- moderate-intensity continuous exercise (Experimental): subjects will exercise at 65% maximal oxygen consumption (VO2max) for 30-45 minutes
  Interventions: Behavioral: Moderate intensity exercise session
- high-intensity interval exercise (Experimental): subjects will completed 10x1minute exercise intervals at maximal oxygen consumption (VO2max) with 1 minute active recovery between
  Interventions: Behavioral: High intensity exercise session

INTERVENTIONS:
Behavioral: Low intensity exercise session — subjects will exercise at 30% maximal oxygen consumption (VO2max) for 45-60 minutes
  Arms: low-intensity continuous exercise
Behavioral: Moderate intensity exercise session — subjects will exercise at 65% maximal oxygen consumption (VO2max) for 30-45 minutes
  Arms: moderate-intensity continuous exercise
Behavioral: High intensity exercise session — subjects will completed 10x1minute exercise intervals at maximal oxygen consumption (VO2max) with 1 minute active recovery between
  Arms: high-intensity interval exercise

SUMMARY:
The study will assess the exercise-induced changes in chromatin accessibility and gene expression in a cell type-specific manner in skeletal muscle from healthy adults in response to exercise at three different intensities - 1) low-intensity continuous exercise, 2) moderate-intensity continuous exercise, and 3) high-intensity interval exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-40
* Body Mass Index: 20-30 kg/m2
* Must engage in regularly planned aerobic-type exercise at moderate-vigorous intensity, 3 times per week for at least 30-60 minutes/session
* Women must have regularly occurring menses and must be premenopausal
* Subject willingness to opt-in for the Michigan Genomics Initiative (MGI) Repository

Exclusion Criteria:

* Evidence/history of cardiovascular or metabolic disease.
* Taking anti-coagulate medications or medications known to affect metabolism or inflammation
* Weight instability ≥ ±3kg in the last 6 months
* Tobacco or e-cigarette users
* Women must not be pregnant or actively lactating

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
post-translational modifications of skeletal muscle oxidative enzymes | 30 minutes before exercise
  Western blot
post-translational modifications of skeletal muscle oxidative enzymes | immediately after exercise
  Western blot
post-translational modifications of skeletal muscle oxidative enzymes | 60 minutes after exercise
  Western blot
post-translational modifications of Adipose tissue metabolic proteins | 15 minutes before exercise
  Western blot
post-translational modifications of Adipose tissue metabolic proteins | 75 minutes after exercise
  Western blot
mRNA expression of skeletal muscle oxidative enzymes | 30 minutes before exercise
  qPCR
mRNA expression of skeletal muscle oxidative enzymes | immediately after exercise
  qPCR
mRNA expression of skeletal muscle oxidative enzymes | 60 minutes after exercise
  qPCR
mRNA expression of adipose tissue metabolic enzymes | 15 minutes before exercise
  qPCR
mRNA expression of adipose tissue metabolic enzymes | 75 minutes after exercise
  qPCR

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States